CLINICAL TRIAL: NCT06115369
Title: Examining the Impact of Medically Tailored Meals vs Produce Supplements Delivered Conditionally vs Not on Health Engagement and Health Outcomes Among Patients With Heart Failure
Brief Title: Food Supplementation Delivered Conditionally vs Not Among Patients With Heart Failure
Acronym: FOOD-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ambarish Pandey, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STU-2023-0978
Record Dates: First submitted 2023-10-24; First posted 2023-11-03 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure
Keywords: Heart Failure; Produce; Medically Tailored Meals; Patient Participation
MeSH Terms: conditions — Heart Failure; Patient Participation

STUDY DESIGN:
Intervention Model Description: The study will be designed as a 2 x 2 factorial randomized clinical trial. First, study patients will be randomized 1:1:1 to receive weekly medically tailored meals (MTM) for twice daily consumption (N = 50) vs. weekly fresh produce box (N = 50) vs. a control arm (usual care with dietary counseling only) (N=50). In the second factorial intervention, participants will be randomized 1:1 to receive their food supplements in a conditional fashion, based on whether they attend clinic visits and fill their medications (N =50) vs. receiving the intervention unconditionally (N =50). The intervention will be initiated within a week of hospital discharge and will continue for a period of 90 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Medically Tailored Meals (Experimental): Season Health, our food intervention partner, will provide participants with weekly deliveries of twice daily prepared medically tailored meals (MTM; 14 total per week). Study participants will be able to select choices for these in conjunction with a dietician. The study team will work with Season Health to create customizations to allow for the incorporation of patient dietary preferences. Study team members will assist patients in setting up their Season Health accounts.
  Interventions: Dietary Supplement: Medically Tailored Meals Delivered Conditionally; Dietary Supplement: Medically Tailored Meals Delivered Unconditionally
- Fresh Produce (Experimental): We will work with Season Health, our food intervention partner to provide participants with weekly deliveries of a large box full of fresh produce and pantry staples. The study participants will be able to select choices for these from a large selection of health options in conjunction with a dietician. The study team will work with Season Health to create customizations to allow for the incorporation of patient dietary preferences. Study team members will assist patients in setting up their Season Health accounts.
  Interventions: Dietary Supplement: Produce Boxes delivered Conditionally; Dietary Supplement: Produce Boxes Delivered Unconditionally
- Control arm (No Intervention): This control arm will receive dietary education only with usual heart failure care.

INTERVENTIONS:
Dietary Supplement: Medically Tailored Meals Delivered Conditionally — Season Health, our food intervention partner, will provide participants with weekly deliveries of twice-daily prepared medically tailored meals (MTM). Participants will receive this supplement conditioned on continued participation and engagement in their healthcare, including attending all scheduled office visits and refilling prescription medications. If participants do not refill their prescriptions or do not attend their office visits, the shipments of medically tailored meals will be paused. These will be restarted when the participant's appointment is rescheduled or when the participant's prescription is refilled.
  Arms: Medically Tailored Meals
Dietary Supplement: Medically Tailored Meals Delivered Unconditionally — Season Health, our food intervention partner, will provide participants with weekly deliveries of twice-daily prepared medically tailored meals (MTM). Participants will receive this supplement unconditionally for the entire study duration.
  Arms: Medically Tailored Meals
Dietary Supplement: Produce Boxes delivered Conditionally — Season Health, our food intervention partner, will provide participants with weekly deliveries of fresh produce and pantry staples. Participants will receive this supplement conditioned on continued participation and engagement in their healthcare, including attending scheduled office visits and refilling prescription medications. If participants do not refill their prescriptions or do not attend their office visits, the shipments of medically tailored meals will be paused. These will be restarted when the participant's appointment is rescheduled or when the participant's prescription is refilled.
  Arms: Fresh Produce
Dietary Supplement: Produce Boxes Delivered Unconditionally — Season Health, our food intervention partner, will provide participants with weekly deliveries of fresh produce and pantry staples. Participants will receive this supplement unconditionally throughout the entire study period.
  Arms: Fresh Produce

SUMMARY:
The current study proposes to investigate if the provision of healthy food can improve outcomes following discharge after HF hospitalization. To investigate this in an efficient and pragmatic manner, a factorial randomized control trial design will be utilized to simultaneously investigate two separate, important food-related questions:

* Does the provision of 90 days of either medically-tailored meals or fresh produce boxes improve 90-day patient outcomes among those with HF relative to a control group not receiving food supplements and instead receiving an equivalent monetary supplement?
* Does receipt of the supplement in a conditional fashion, where the supplement is continued only if the participant attends follow-up visits or fills prescribed medications at the pharmacy, have more impact than providing unconditional supplementation?

DETAILED DESCRIPTION:
Eating a nutritious diet is important for maintaining health. However, getting healthy foods can be a challenge for many individuals whose food shopping is limited by finances, location, or physical limitations from pre-existing health problems. For such in-need individuals, providing supplemental healthy meals can improve their diet and potentially improve their health outcomes. Additionally, getting food supplements can also be a powerful incentive to encourage healthy behaviors.

Individuals with heart failure (HF) present a unique population to assess the value of food supplementation both for its nutritional value and as a health engagement incentive. HF is a common, high-cost public health problem in the United States. Hospitalizations for HF are associated with high rates of mortality, readmission, worsened quality of life, and burgeoning healthcare expenditures. During the post-discharge period, patients are exceptionally vulnerable to a wide variety of adverse health events due to multi-system physiologic impairments. Roughly 20% of all patients with Medicare are readmitted within 30 days, and many are readmitted for different causes than the principal diagnosis of the index admission. While multifactorial, frequent contributing causes of HF readmission include dietary indiscretion, failure to take medications, and failure to follow up with healthcare providers.

Prior studies demonstrate that patients with HF often have food insecurity and non-ideal diets. Nationally, food insecurity among those patients with cardiovascular diseases has increased. Those with HF specifically had some of the highest rates of food insecurity, and the prevalence of food insecurity rose from 11.3% in 1999-2000 to 45.3% in 2017-2018.

Studies have also investigated whether providing food supplements to patients with HF can potentially also improve health outcomes. In a recent cohort study, Medicare Advantage patients with acute heart failure (HF) were given up to 4 weeks of post-hospitalization home-delivered meals. Compared with historical controls, those receiving these meals were significantly less likely to have all-cause readmission and death. In contrast, a recent randomized clinical trial found that providing 10 weeks of medically tailored meals to patients with chronic diseases hospitalized during the COVID-19 pandemic did not lead to reductions in risk of 90-day readmission. However, in an exploratory sub-analysis, patients with HF who had the medically tailored meal intervention had significant reductions in readmissions. While these data are supportive of the hypothesis, they are not definitive, and a prospective randomized trial among patients with HF is needed to rigorously support the efficacy of food support in the post-discharge period to reduce readmission. There is also limited information on the type and means of food supplementation may affect its efficacy.

Based on this background, the current study proposes to investigate if the provision of healthy food can improve outcomes following discharge after HF hospitalization. To investigate this in an efficient and pragmatic manner, a factorial randomized control trial design will be used that will simultaneously investigate two separate important food-related questions. The first factorial design question will evaluate the direct impact of two nutritional supplementation strategies on rehospitalizations and ED visits for HF. Specifically, those hospitalized for HF will be randomized at hospital discharge to either 90 days of healthy medically tailored full meals (MTM) (n=50) or 90 days of a weekly fresh produce box (n=50) or to a control arm (usual care receiving no food supplements with dietary education only) (N=50).

The second factorial intervention will determine whether food supplements can be used as an incentive to increase patient engagement in their own care (i.e., attending a follow-up clinic visit and filling their prescriptions). Specifically, participants receiving food supplementation will be randomized 1:1 to receive their food supplements (MTMs or produce box) in an unconditional or conditional fashion based on the participant successfully attending their clinic visits and filling their medication.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 18 years age with a recent hospitalization for acute decompensated HF

Exclusion Criteria:

* Baseline hyperkalemia with K > 5.5 mEq/L or history of hyperkalemia requiring hospitalization for urgent treatment,
* Receipt of a heart transplant or left ventricular assist device,
* Use of inotropic therapy at hospital discharge,
* Discharge to a skilled nursing facility or long-term care facility that provides prepared patient meals, comorbidity with expected survival < 6 months, and
* Inability to provide an address to receive produce shipments (including unhoused individuals or individuals residing in temporary housing shelters).
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with a readmission or emergency department visit for HF | 90 days
  Total readmissions or visits to the emergency department for HF

SECONDARY OUTCOMES:
Hierarchical Composite Endpoint | 90 days
  Win-ratio based endpoint with the following hierarchy: (1) mortality, (2) readmission or ED visit for HF (total), (3) ≥10 point improvement in Kansas City Cardiomyopathy Questionnaire (KCCQ) - Clinical Summary Score (CSS). The KCCQ clinical summary score ranges from 0 to 100, where higher scores indicating better quality of life.
Between group change in Kansas City Cardiomyopathy Questionnaire - Clinical Summary Score | The survey will be assessed at baseline and at 90 days at the conclusion of the study.
  The KCCQ clinical summary score ranges from 0 to 100, where higher scores indicating better quality of life.
Medication adherence | 90 days
  Morisky Medication Adherence Score. Scores are summed from 0 to 8, with higher scores meaning better adherence.
Attendance to scheduled clinic appointments | 90 days
  Percent from 0-100%, calculated by the number of attended visits divided by the number of scheduled visits after excluding cancelled visits (either cancelled by provider or participant)
Filling of outpatient medication prescription | 90 days
  Percent from 0-100%, calculated by percent of new prescriptions filled at pharmacy divided by number of prescriptions sent to pharmacy by providers

CONTACTS AND LOCATIONS:
Overall Officials: Ambarish Pandey, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No